CLINICAL TRIAL: NCT02875158
Title: Modified Settings for Transscleral Cyclophotocoagulation of the Ciliary Body in Glaucoma : A Randomized Controlled Trial
Brief Title: Cyclophotocoagulation in Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-2212
Record Dates: First submitted 2016-07-18; First posted 2016-08-23 (Estimated); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diode laser using conventional settings (Active Comparator): The cyclophotocoagulation protocol is used with the conventional cyclophotocoagulation settings of 2000 mW for 2 seconds.
  Interventions: Procedure: Cyclophotocoagulation protocol; Procedure: Conventional cyclophotocoagulation
- Diode laser using modified settings (Experimental): The cyclophotocoagulation protocol is used with the modified cyclophotocoagulation settings of 1250 mW for 4 seconds.
  Interventions: Procedure: Cyclophotocoagulation protocol; Procedure: Modified cyclophotocoagulation

INTERVENTIONS:
Procedure: Cyclophotocoagulation protocol — * Intravenous route is installed
  * Retrobulbar anaesthesia : 50% xylocaine (2%) + 50% bupivicaine
  * Parameters set for laser treatment (1250mW-4seconds or 2000mW-2 seconds depending on the assigned group)
  * Pars plana measurement using transillumination (if needed)
  * Laser treatment applied approximately 1mm post to limbus
  * Dexamethasone 0,5 mg subconjunctival injection
  * Post-op regimen: Prednisolone 1% qid x 4 weeks, Atropine 1% bid x 2 weeks + Erythromycin ointment + patch x 6h
Procedure: Conventional cyclophotocoagulation — 1250 mW for 4 seconds.
  Arms: Diode laser using conventional settings
Procedure: Modified cyclophotocoagulation — 2000 mW for 2 seconds.
  Arms: Diode laser using modified settings

SUMMARY:
Transscleral cyclophotocoagulation of the ciliary body is an effective technique to reduce intraocular pressure in case of glaucoma. Due to concerns over complications, the main indications for this second-line treatment are refractory glaucoma medication / surgery and low visual prognosis. The 2000 milliwatts (mW) for 2 seconds settings are used by the majority of researchers and clinicians according to the published literature. Some have proposed using 1250 mW for 4 seconds to improve the use of this medical procedure.

The aim of this study is to determine how different parameters affect the efficacy of the treatment. This is a prospective double-blinded randomized controlled trial comparing two groups, the experimental group using 1250 mW for 4 seconds and the control group using 2000 mW for 2 seconds.

ELIGIBILITY:
Inclusion Criteria:

* Patients with poorly controlled high pressure glaucoma
* Cyclophotocoagulation necessary to prevent visual loss
* Cyclophotocoagulation necessary to prevent or to reduce ocular discomfort

Exclusion Criteria:

* Patient has already undergone a cyclophotocoagulation or cryotherapy treatment in the same eye for glaucoma
* Patients receiving concomitant treatment the same day as the intervention
* Patient not able to follow the prescribed post-operative treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) evolution | 1h, 1 month, 6 months, 12 months, 18 months and 24 months post-op
  The intraocular pressure is measured to determine the efficacy of treatment during follow-up compared to the baseline IOP.

SECONDARY OUTCOMES:
Presence of complications | During the intervention, 1 month, 6 months, 12 months, 18 months, 24 months post-op
  Assessment of complications (if applicable).
Use of medication | 1 month, 6 months, 12 months, 18 months and 24 months post-op
  Assessment of the topical and oral glaucoma medication at baseline and after treatment
Retreatment | From the initial treatment up to the last visit (24 months)
  The clinician will assess the need for retreatment based on clinical experience.
Visual acuity | 1 month, 6 months, 12 months, 18 months and 24 months post-op
  The visual acuity will be assessed at baseline and each subsequent visit

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Toren, Doctor, Principal Investigator — Centre de recherche du CHU de Québec : Université Laval
Locations (1):
- Centre universitaire d'ophtalmologie, Hôpital du Saint-Sacrement. CHU de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No